CLINICAL TRIAL: NCT01823848
Title: A Randomized Controlled Trial of Three Types of Enemas Used to Treat Functional Constipation in Children
Brief Title: A Trial of Three Types of Enemas Used to Treat Functional Constipation in Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Ara Festekjian, Assistant Professor of Clinical Pediatrics, Children's Hospital Los Angeles
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CCI-12-00295
Record Dates: First submitted 2013-03-26; First posted 2013-04-04 (Estimated); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Functional Constipation
Keywords: constipation; enema
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sodium phosphate enema (Active Comparator): Administration of sodium phosphate (fleets) enema for functional constipation in children ages 4-12 years Age 4-5: 33ml per rectum Age 5-12: 66ml per rectum
  Interventions: Drug: Sodium phosphate enema; Drug: Normal saline enema; Drug: Mineral oil enema
- Normal saline enema (Active Comparator): Administration of normal saline enema for functional constipation in children ages 4-12 years Admininstered as 10ml/kg with maximum of 700ml
  Interventions: Drug: Sodium phosphate enema; Drug: Normal saline enema; Drug: Mineral oil enema
- Mineral oil enema (Experimental): Administration of mineral oil enema for functional constipation in children ages 4-12 years Administered as 66ml per rectum
  Interventions: Drug: Sodium phosphate enema; Drug: Normal saline enema; Drug: Mineral oil enema

INTERVENTIONS:
Drug: Sodium phosphate enema — Rectally administered medication to treat constipation
  Other Names: Fleets enema
Drug: Normal saline enema — Rectally administered medication to treat constipation
Drug: Mineral oil enema — Mineral oil enema administered to treat constipation. 66ml per rectum

SUMMARY:
Functional constipation is extremely common in children and is defined as painful, hard stools or firm stools for twice or less per week. Functional constipation accounts for 3% of general pediatric visits and up to 25% of pediatric gastroenterology visits. Constipation and fecal impaction can lead to a range of symptoms including decreased appetite, vomiting, and abdominal pain frequently resulting in Emergency Department (ED) presentation. In contrast to the outpatient setting where diet and oral medications work well to relieve symptoms related to functional constipation, ED management requires an approach with quicker results. For immediate relief of symptoms, disimpaction via enema use may be better than polyethylene glycol (PEG) 3350 for children. However, the type of enema to be used is not well studied. Currently, any patient presenting to the ED with a presumed diagnosis of abdominal pain due to functional constipation receives an oral dose of PEG and one of the following three types of enemas (based on the ED treating attending's discretion): phosphate or Fleets enema, normal saline enema, or mineral oil enema. There is no evidence in the literature that demonstrates any difference in the effectiveness of each of these enemas. The investigators propose a randomized control trial of the three types of pediatric enemas readily used in our ED to determine the best approach. There will be three arms within this study: a) PEG plus phosphate enema b) PEG plus normal saline enema and c) PEG plus mineral oil enema. The physicians enrolling patients will not be the treating physicians. The four principal investigators (blinded to the type of enema being used), following appropriate informed consent, will obtain pain scores (Faces Pain Scale - Revised) pre- and post-administration of each of the three treatments listed above in order to determine the best enema to use in children 4-12 years of age. Other outcomes to be analyzed will include the patient's weight pre- and post-administration of the enema, satisfaction ratings on a visual analog scale from the treating physician (who will also be blinded), and parental surveys on the day of administration and 3-5 days following discharge. Data analysis for pain scores will be completed with repeated measures anova. Categorical values will be compared using Chi Square analysis and continuous variables will be compared using parametric statistics.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-12 years
* Receiving enema in ED for presumed constipation

Exclusion Criteria:

* Critically ill patient
* Any history of renal insufficiency, renal disease, or elevated creatinine
* Any history of intestinal anatomic abnormality (i.e. anal stenosis, anal surgery, bowel obstruction, hirschprung's disease)
* An inability to self-report pain
* Presence of gastrostomy or jejunostomy tube
* Any history of gastrointestinal dysmotility
* Inability to read or speak English or Spanish

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2013-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in pain scores following administration of enema | 1-2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ara Festekjian, MD, Principal Investigator — CHLA Division of Emergency Medicine
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No